CLINICAL TRIAL: NCT01078441
Title: A Phase II Study of Bortezomib, Liposomal Doxorubicin, Dexamethasone, and Cyclophosphamide in Patients With Multiple Myeloma Relapsing Within 12 Months of Autologous Stem Cell Transplant
Brief Title: Bortezomib, Liposomal Doxorubicin Hydrochloride, Dexamethasone, and Cyclophosphamide in Treating Patients With Multiple Myeloma That Relapsed After Autologous Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed early due to weak accrual on June 26, 2012.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02002; NCI-2011-02002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E2A08 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2010-02-27; First posted 2010-03-02 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-07

CONDITIONS: Refractory Multiple Myeloma
Keywords: Bortezomib; Liposomal Doxorubicin; Dexamethasone; Cyclophosphamide; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — liposomal doxorubicin; Bortezomib; Dexamethasone; Calcium Dobesilate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive bortezomib 1.3 mg/m2 subcutaneously on days 1, 8, and 15; liposomal doxorubicin 30 mg/m2 intravenously (IV) over 1 hour on day 4; oral dexamethasone 20mg on days 1, 2, 8, 9, 15 and 16; and cyclophosphamide 750 mg/m2 IV over 2 hours on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: liposomal doxorubicin; Drug: bortezomib; Drug: dexamethasone; Drug: cyclophosphamide

INTERVENTIONS:
Drug: liposomal doxorubicin — Given IV
  Other Names: Doxil; Doxorubicin HCl Liposomal; Doxorubicin Hydrochloride Liposomal; Doxorubicin Hydrochloride Liposome
Drug: bortezomib — Given subcutaneously.
  Other Names: Velcade; PS-341; MLN-341; LDP-341
Drug: dexamethasone — Given orally
  Other Names: Decadron; Hexadrol; Dexameth; Dexone; DXM
Drug: cyclophosphamide — Given IV
  Other Names: CTX; Cytoxan; Neosar

SUMMARY:
This phase II trial is studying how well giving bortezomib together with liposomal doxorubicin hydrochloride, dexamethasone, and cyclophosphamide works in treating patients with multiple myeloma that relapsed after autologous stem cell transplant. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as liposomal doxorubicin hydrochloride, dexamethasone, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with liposomal doxorubicin hydrochloride, dexamethasone, and cyclophosphamide may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 1-year survival of patients with relapsed multiple myeloma treated with bortezomib, liposomal doxorubicin, dexamethasone, and cyclophosphamide.

SECONDARY OBJECTIVES:

I. To evaluate response rates in patients treated with this regimen.

II. To evaluate the median time to progression in patients treated with this regimen.

III. To evaluate the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive bortezomib 1.3 mg/m2 subcutaneously on days 1, 8, and 15; liposomal doxorubicin 30 mg/m2 intravenously (IV) over 1 hour on day 4; oral dexamethasone 20mg on days 1, 2, 8, 9, 15 and 16; and cyclophosphamide 750 mg/m2 IV over 2 hours on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

Peripheral blood and bone marrow samples may be collected for future research. Patients complete the Functional Assessment of Cancer Therapy (FACT) neurotoxicity questionnaire periodically.

After completion of study treatment, patients are followed up every 3 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma that was symptomatic at the time of initial diagnosis
* Must have met the following criteria at one point during the disease course:

  * Bone marrow plasmacytosis with ≥ 10% plasma cells or sheets of plasma cells or biopsy-proven plasmacytoma
  * Symptomatic disease at initial diagnosis that prompted the initiation of therapy as well as evidence of end-organ damage at the time of diagnosis, including at least 1 of the following:

    * Anemia
    * Hypercalcemia
    * Bone disease (lytic bone lesions or pathologic fracture)
    * Renal dysfunction
* Disease relapsed < 12 months after autologous stem cell transplantation (SCT)
* Measurable disease, as defined by the presence of ≥ 1 of the following:

  * Serum M-spike ≥ 1 g/dL
  * Urine M-spike ≥ 200 mg/24 hours
  * Involved free light chain (FLC) ≥ 10 mg/dL (provided the serum FLC is abnormal)
  * Plasma cells ≥ 30%
* ECOG performance status 0-2
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 14 days since prior palliative and/or localized radiotherapy
* Left ventricular ejection fraction (LVEF) normal by Echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan
* Hemoglobin > 8 g/dL
* Platelet count ≥ 75,000/mm^3 (without transfusion support)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (without use of growth factors)
* Creatinine < 2.5 mg/dL
* Direct bilirubin ≤ 1.5 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal
* All tests below must be performed within 14 days prior to registration:

  * Serum free light chain assay
  * Kappa free light chain
  * Lambda free light chain
* Prior malignancy allowed provided it was treated curatively and has not relapsed in 5 years

  * Patients with basal cell skin cancer, in situ cervical cancer, or prostate cancer not requiring therapy are eligible

Exclusion Criteria:

* Therapy for relapsed disease following SCT
* Known allergy to bortezomib or anthracyclines
* Prior allogeneic SCT
* Peripheral neuropathy ≥ grade 2 according to the Cancer Therapy Evaluation Program (CTEP) active version of the NCI Common Terminology Criteria for Adverse Events (CTCAE)
* Concurrent uncontrolled illness that would limit study compliance, including the following:

  * Uncontrolled hypertension
  * Symptomatic congestive heart failure
  * Unstable angina
  * Uncontrolled cardiac arrhythmia
  * Uncontrolled psychiatric illness or social situation
  * Active uncontrolled infection
* Prior doxorubicin hydrochloride exposure > 240 mg/m^2
* Active, uncontrolled seizure disorder
* Seizures within the past 6 months
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, M.D., Study Chair — Mayo Clinic
Locations (130):
- United States (130):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Medical Center of Central Georgia, Macon, Georgia
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Union Hospital of Cecil County, Elkton MD, Maryland
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Community Health Partners Regional Medical Center, Elyria, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Butler Memorial Hospital, Butler, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two patients were enrolled from ECOG member institutions between September 14, 2010 and June 26, 2012. The study was closed early due to weak accrual.
Groups:
- Treatment (Combination Chemotherapy): Patients receive bortezomib subcutaneously on days 1, 8, and 15; liposomal doxorubicin intravenously (IV) over 1 hour on day 4; oral dexamethasone on days 1, 2, 8, 9, 15 and 16; and cyclophosphamide IV over 2 hours on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  liposomal doxorubicin: Given IV
  bortezomib: Given subcutaneously.
  dexamethasone: Given orally
  cyclophosphamide: Given IV
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled are included in this analysis.
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 51 [48 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: One-year Survival in Patients Treated With This Regimen.
Description: Proportion of patients who are still alive at 1 year after registration.
Time Frame: Assessed at 1 year
Population: All eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of patients
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 2
Proportion of patients | 0.5 [0.03 to 0.97]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Combination Chemotherapy: Patients receive bortezomib subcutaneously on days 1, 8, and 15; liposomal doxorubicin intravenously (IV) over 1 hour on day 4; oral dexamethasone on days 1, 2, 8, 9, 15 and 16; and cyclophosphamide IV over 2 hours on day 1. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Chemotherapy (N=2)
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Chemotherapy (N=2)
Anemia (Blood and lymphatic system disorders) | 1
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less